CLINICAL TRIAL: NCT03481933
Title: Investigation of the Therapeutic Value of Transcranial Stimulation With Direct Current on Language Disorders in Semantic Dementia
Brief Title: Evaluation of a Transcranial Stimulation With Direct Current on Language Disorders in Semantic Dementia
Acronym: STIM-SD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P160937J
Record Dates: First submitted 2018-03-09; First posted 2018-03-29 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2023-03

CONDITIONS: Semantic Dementia
MeSH Terms: conditions — Frontotemporal Dementia

STUDY DESIGN:
Intervention Model Description: left-excitatory tDCS ; right-inhibitory tDCS; sham tDCS (placebo)
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1:left-excitatory tDCS (Experimental): 20 SD patients who receive left-excitatory trans cranial stimulation
  Interventions: Device: Transcranial stimulation
- 2:right-inhibitory tDCS (Active Comparator): 20 SD patients who receive right-inhibotory trans cranial stimulation
  Interventions: Device: Transcranial stimulation
- 3:sham tDCS (Sham Comparator): 20 SD patients who receive sham stimulation
  Interventions: Device: Transcranial stimulation

INTERVENTIONS:
Device: Transcranial stimulation — 1. 10 days of stimulation (20min, 1.59mA) in double-blind sham-controlled. 3 arms (N=20 in each arm):
     * left-excitatory tDCS (N=20)
     * right-inhibitory tDCS (N=20)
     * sham tDCS (N=20)
  2. 4 language/semantic evaluations: base-line; 3 days; 2 weeks; 4 months post-tDCS
  3. 2 MRI/PET acquisitions: pre-stimulation (base-line); 2 weeks post-tDCS

SUMMARY:
Within the spectrum of fronto-temporal lobar degeneration (FTLD) semantic dementia (SD) causes profound language dysfunction. SD damages semantic processing typically in the temporal poles (anterior temporal lobes, ATL). It is an early onset disease (often before 65 years of age) affecting about 4000 patients in France and for which no validated treatment is available.

For several years a growing number of studies have explored the effects of transcranial stimulation (TCS) on aphasic patients following stroke. Several studies have targeted left-sided language areas and/or homotopical right-sided regions with excitatory or inhibitory TCS, respectively, according to the principle of inter-hemispheric inhibition. In addition, repetitive multi-day TCS has provided evidence for long-lasting language effects (>6 months) presumably linked to stimulation-induced neuroplasticity. Such investigations have provided promising results and have demonstrated that the stimulation site is a determining factor by showing that stimulation of cortical areas belonging to the language network usually results in more convincing effects than stimulating areas outside that network. Despite these findings the use of TCS in degenerative language diseases, such as primary progressive aphasias including SD, has only been explored in few small cohort studies and, surprisingly, they have not targeted language-related cortices.

This project proposes the application of multi-day repetitive TCS with direct current (tDCS) in a large population of SD patients (N=60). It is built on a exploratory investigation of our team which has used three single tDCS sessions in a double-blind sham-controlled study. Excitatory and inhibitory tDCS to the left and right temporal pole, respectively, demonstrated highly significant transient effects (20 min) on semantic processing in 12 SD patients, providing 'proof of concept' and the rationale for this project. The aim here consists of using repetitive multi-day tDCS for a potential therapeutic outcome leading to long-lasting semantic improvement via neuroplasticity. The project is grounded on 2 hypotheses: i) tDCS to temporal poles (left-excitatory, right-inhibitory) reactivates semantic processing in SD, ii) repetitive tDCS during ten days could induce neuroplasticity and therapeutic language improvement.

DETAILED DESCRIPTION:
Main objective and evaluation criteria:

To evaluate the potential therapeutic efficacy of repetitive tDCS during 10 days on language/semantic impairment in SD via a double-blind sham-controlled study design. The evaluation criteria will be a significant improvement of language/semantic performances two weeks after tDCS as compared to base-line (before tDCS), contrasting subgroups receiving left-excitatory or right-inhibitory tDCS vs. sham tDCS

Secondary objectives and evaluation criteria:

1. Assess the time course of potential language/semantic improvement through the application of four follow-up time-points: base-line (max one week before tDCS), three days, two weeks and four months after tDCS. The evaluation criteria will be significant improvement/modulation of language/semantic performances, comparing performances at the four time-points.
2. Assess brain markers which could reflect stimulation-induced neuroplasticity. Evaluation criteria will be significant modulation of cortical metabolism (FDG-PET) and functional connectivity (fMRI resting-state) comparing base-line and the 'two-week' time-point.
3. Compare left-excitatory and right-inhibitory tDCS to reveal the most efficient stimulation modality. Evaluation criteria will be a detection of a potential outcome difference between left-excitatory and right-inhibitory tDCS on the performance within the different language/semantic tasks.
4. Improve the understanding of the semantic roles of the left and right temporal pole, and their potential anatomical connectivity, by comparing left and right temporal pole stimulation and using MRI-based fiber tracking. 4) Improve the understanding of the semantic roles of the left and right temporal pole, and their potential anatomical connectivity, by comparing left and right temporal pole stimulation and using MRI-based fiber tracking.

Experimental design :

10 days of stimulation (20min, 2mA). Four language/semantic evaluations: base-line; 3 days; 2 weeks; 4 months post-tDCS. Two MRI/PET acquisitions: pre-stimulation (base-line); 2 weeks post-tDCS

Population :

Patients with semantic dementia (SD). Healthy controls for normative measures (no tDCS for controls)

Testing treatment :

tDCS (specific device) : NE STARSTIM-ENOBIO 8 channels.

Practical procedure :

The duration of the study will be 41 months; 36 months being dedicated to patient inclusion. Participation duration of a patient will be of 4 months and 1 week to 4 months and 3 weeks maximum. First, patients will undergo a series of standardized neuropsychological and language tests that are included in routine care and inclusion criteria will be checked. After inclusion, the base-line visit will comprehend 1) MRI/PET in the Nuclear Medicine Service (CHU Pitié Salpêtrière), and 2) language/semantic tasks at the Department of Neurology (CHU Pitié Salpêtrière). Subsequently the ten stimulation sessions will be scheduled. They will take place in the Institute of Memory and Alzheimer's disease (Department of Neurology, CHU Pitié Salpêtrière) during two consecutive weeks (20 minutes of tDCS). The tDCS sessions will be followed by three time-point visits: 3 days (time-point 2) and two weeks (time-point 3) after the last stimulation session patients will undergo the language/semantic tasks. At time point 3 the second MRI/PET acquisition will take place. Finally, the visit of time-point 4 will be at four months after the last tDCS session, dedicated to a last application of language/semantic tasks.

Selected number of subjects:

80 SD patients selected in order to have 60 randomized into three arms (20 patients/arm).Two arms receiving active tDCS versus one receiving sham tDCS.

20 healthy volunteers will be included (participants will provide normative language/semantic scores and MRI/PET measures; they will not undergotDCS).

Number of centers: 3 centers in France (Paris)

Research duration:

Inclusion period: 36 months Participation period (Selection/inclusion, tDCS sessions and evaluation at 4 time-points): 4 months and 1 week to 4 months and 3 weeks Total duration: 41 months

Funding source: AP-HP (Assistance Publique des Hôpitaux de Paris).

ELIGIBILITY:
Inclusion Criteria:

SD-Patients:

1. Patients fulfilling the international diagnosis criteria of SD (Gorno-Tempini et al., 2011): fluent speech, single word comprehension and naming deficit, +/- object recognition deficits, +/- surface agraphia or alexia. Absence of phonemic paraphasias, agrammatism and word apraxia.
2. Age > 18 years old.
3. Patients have given their informed written consent.
4. Affiliation to a social security regime.

Healthy controls:

1. Age >18 years old
2. Subjects have given their informed written consent.
3. Subjects selected according to the matching criteria (age, sex, handedness and number of years of education).
4. Affiliation to a social security regime

Exclusion Criteria:

SD-Patients:

1. MADRS ≥ 20 (major depressive syndrome according to the DSM-IV-R criteria)
2. MMS < 10/30
3. FAB < 7/18
4. BDAE aphasia severity rating scale < 3/5
5. Patients not having French as their mother tongue
6. Other neurological pathology or general disorder or major physical deficits than can interfere with cognitive functioning
7. MRI or PET contraindication, 18-FDG contraindication
8. Cerebral MRI data compatible with a pathological process other than the one related to SD (Vascular, traumatic, tumoral, infectious, or metabolic brain injury). A moderate or discrete leukoaraiosis will not be considered as a non- inclusion criterion (patients with a Fazekas and Schmidt [Fazekas et al., 1998a; fazekas et al., 1998b],stage >2 for hypersignals of the periventricular and deep white matter will not be included)
9. The patient should not participate simultaneously in another brain therapeutic trial (possibility of bias between stimulation and evaluation of the effect on language / semantic processes)
10. - tDCS contraindications: epilepsy antecedents, presence of epilepsy risk factors (known alcoholism or metabolic troubles, antecedents of head injury or chirurgical intervention on the brain or the skull), skin lesions of the scalp, skull metal implants.
11. - Patients under curatorship or tutorship
12. - Women whose pregnancy is known or who do not have effective contraception if they are of reproductive age (checked by urinary test), breastfeeding.

Healthy controls:

1. Subjects not having French as their mother tongue
2. Subjects having a neurological or psychiatric disease or major deficits than can interfere with cognitive functioning
3. MRI or PET contraindication, 18-FDG contraindication
4. Women whose pregnancy is known or who do not have effective contraception if they are of reproductive age (checked by urinary test), breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-05-16 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Significant improvement of semantic performances on the experimental 'semantic matching test' | 15 days
  The 'semantic matching test' assesses semantic processing in the verbal and visual modality. Outcome measure will be the difference between performance on the test at base line and two weeks after tDCS: composite score of accuracy on the test.

SECONDARY OUTCOMES:
Significant modulation of semantic performances on the 'semantic matching test' | 3 days, 4 months
  Outcome measures will be the difference of performance on the test between base line and 1) 3 days after tDCS, 2) 4 months after tDCS: composite score of accuracy on the test.
significant modulation of cortical metabolism and functional connectivity | 2 weeks
  significant modulation of cortical metabolism on FDG-PET and functional connectivity on fMRI resting-state, comparing base-line and the two weeks after tDCS
Detection of a potential outcome difference between left-excitatory and right-inhibitory tDCS | 15 days, 4 months
  performance difference on the accuracy score of the semantic matching task comparing left and right tDCS

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Département de Neurologie - Centre des maladies neurologiques, cognitives et comportementales, Paris
  - Hôpital de la Pitié-Salpétrière, Paris

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sanches C, Levy R, Benisty S, Volpe-Gillot L, Habert MO, Kas A, Stroer S, Pyatigorskaya N, Kaglik A, Bourbon A, Dubois B, Migliaccio R, Valero-Cabre A, Teichmann M. Testing the therapeutic effects of transcranial direct current stimulation (tDCS) in semantic dementia: a double blind, sham controlled, randomized clinical trial. Trials. 2019 Nov 20;20(1):632. doi: 10.1186/s13063-019-3613-z. PMID 31747967